CLINICAL TRIAL: NCT04460924
Title: ARTiBIOME: Effect of HIV and ART on Gut Microbiome
Brief Title: ARTiBIOME: Observational Study on the Effect of HIV and ART on Gut Microbiome
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ARTiBIOME: Observational study
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- MSM HIV-uninfected and ART naïve: Men who have sex with men without HIV infection, not receiving ART
- MSM HIV-infected starting ART: Men who have sex with men with HIV infection, starting ART
  Interventions: Drug: Integrase strand transfer inhibitors
- MSM HIV-infected on ART with >500 CD4 Tcells: Men who have sex with men with HIV infection, on ART and with >500 CD4 T cells/uL
  Interventions: Drug: Integrase strand transfer inhibitors
- MSM HIV-infected on ART with <350 CD4 Tcells: Men who have sex with men with HIV infection, on ART and with <350 CD4 T cells/uL
  Interventions: Drug: Integrase strand transfer inhibitors
- MSM HIV negative patients starting PEP with INST: Men who have sex with men without HIV infection, starting post-exposure prophylaxis with raltegravir
  Interventions: Drug: Integrase strand transfer inhibitors

INTERVENTIONS:
Drug: Integrase strand transfer inhibitors — Integrase strand transfer inhibitors as post-exposure prophylaxis or as antiretroviral treatment
  Groups: MSM HIV negative patients starting PEP with INST; MSM HIV-infected on ART with <350 CD4 Tcells; MSM HIV-infected on ART with >500 CD4 Tcells; MSM HIV-infected starting ART

SUMMARY:
Antiretroviral treatment for HIV has allowed patients to have undetectable viral load indefinitely. Despite that, HIV infection has become a chronic inflammatory disease, with increased mortality. This pro-inflammatory state is in part explained by the dysbiosis of intestinal bacterial populations. However, little is known on the impact of the antiretroviral treatment on this population and very few studies have evaluated these alterations.

The aim of this study is to study microbiome on healthy patients and HIV-infected patients exposed to antiretroviral treatment with integrase strand transfer inhibitors.

ELIGIBILITY:
Inclusion criteria:

* Willing to sign consent form
* Men with an age >18 years
* Engagement in insertive or receptive anal intercourse with another men

  *Exclusion criteria:
* Previous history of ART exposure
* Use of antibiotics in the past 3 months
* Previous history of inflammatory bowel disease, autoimmune disease or cirrhosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: We will compare 20 MSM HIV negative patients starting PEP with INSTI with:
  * 20 MSM HIV-uninfected and ART naïve (A)
  * 20 MSM HIV-infected starting ART (B)
  * 20 MSM HIV-infected on ART with >500 CD4 Tcells ( C )
  * 20 MSM HIV-infected on ART with <350 CD4 Tcells (D) (the study population has been restricted to MSM given the strong influence of sexual orientation on the microbiota composition
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Alpha diversity changes of fecal microbiota composition | Baseline and 1 month, 3 months, 12 months
  Alpha diversity changes of fecal microbiota composition between study groups
Beta diversity changes of fecal microbiota composition | Baseline and 1 month, 3 months, 12 months
  Beta diversity changes of fecal microbiota composition between study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal and Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No